CLINICAL TRIAL: NCT06494631
Title: Clinical Study to Assess the Safety and Performance of the Xeltis Hemodialysis Access Graft
Brief Title: Xeltis Hemodialysis Access Graft (aXess) US Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-12
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- aXess graft (Experimental)
  Interventions: Device: Xeltis Hemodialysis Access (aXess) graft

INTERVENTIONS:
Device: Xeltis Hemodialysis Access (aXess) graft — The aXess graft is a sterile, restorative biodegradable polymer-based vascular graft, consisting of a tubular structure with a 6mm inner diameter. It is comprised of a highly porous polymer matrix and an embedded electropolished nitinol reinforcement layer (Strain Relief System). The aXess graft is able to support both straight and loop configurations and may be implanted in the upper arm and forearm.

SUMMARY:
A multi-center, prospective, single-arm, non-randomized, staged, pivotal clinical study to evaluate the safety and performance of the aXess graft in subjects aged 18 and above, diagnosed with end-stage kidney disease, and possessing an estimated glomerular filtration rate (eGFR) less than 20 ml/min, who intend to undergo hemodialysis but are considered unsuitable candidates for fistula creation by the investigating surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with end-stage renal disease (ESRD) who require placement of an AVG in the upper extremity to start (within the first 6 months of follow-up) or maintain hemodialysis therapy and are deemed unsuitable for fistula creation by the investigational surgeon.
2. At least 18 years of age at screening.
3. Suitable anatomy (e.g. a target vein with a minimum diameter of 4mm) for the implantation of an aXess graft
4. The patient has been informed about the nature of the study, agrees to its provisions, and has provided written informed consent.
5. The patient has been informed and agrees to pre- and post-procedure follow-up.
6. Life expectancy of at least 12 months.

Exclusion Criteria:

1. History or evidence of severe cardiac disease (NYHA Functional Class IV and/or EF <25%), myocardial infarction within 6 months of study enrolment, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina.
2. Uncontrolled or poorly controlled diabetes in the opinion of the investigator. Recommended standards of A1c level <8% / 183 mg/dl / 10.2 eAG.
3. Abnormal blood values (e.g., leukopenia with white blood cell count (WBC) <4,000/mm³ and/or anemia with Hemoglobin <8g/dL and/or thrombocytopenia <100,000/mm³) that could influence patient recovery and or/ graft hemostasis.
4. Reduced liver function, defined as: >2x the upper limit of normal for serum bilirubin, International Normalized Ratio (INR) >1.5 or prothrombin time (PT) >18 seconds.
5. Any active local or systemic infection.
6. Known heparin-induced thrombocytopenia.
7. Known active bleeding disorder and/or any coagulopathy or thromboembolic disease.
8. Allergies to study device (nitinol) or agents/medication, such as contrast agents or aspirin, that can't be controlled medically.
9. Anticipated renal transplant within 6 months.
10. Known or suspected central vein obstruction on the side of planned graft implantation.
11. Previous dialysis access graft in the operative limb, unless the aXess graft can be placed more proximally than the previously failed graft.
12. Previous enrollment in this study.
13. Subject is participating in another study.
14. A female who is breastfeeding or of childbearing potential with a positive pregnancy test or not using adequate contraception.
15. Any other condition which, in the judgment of the investigator, would preclude adequate evaluation for the safety and performance of the study conduit.

Intra-operative exclusion criteria:

1. Unsuitable anatomy to implant the aXess graft (e.g., target vein and/or artery diameter not suitable; severe calcification).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Secondary patency rate in survivors | 12 months
  Secondary patency is defined as the interval between vascular access creation and abandonment with or without interventions (operative or endovascular) aimed to maintain or restore the vascular access's functionality.
  Patients who died or changed dialysis modality before 12 months will be excluded from the primary effectiveness analysis if loss of secondary patency was not observed before these events
Rate of device related infections and bleeding | 12 months
  Infections are defined as: All device or procedure related infections potentially resulting from surgical manipulations or device cannulation, including both minor and major infections., Bleeding (procedure or device related bleeding, at least BARC 2) and device related hematoma defined as blood accumulation around the graft arising from the implantation or cannulation that triggered a medical or surgical action

SECONDARY OUTCOMES:
Freedom from device-related SAE | Discharge, 1, 3, 6, 12, 18, 24, and 60 months
Implantation success rate | 1 day, from moment of implant until discharge
  Defined as a technically successful aXess graft implantation in the planned configuration, free from kinking and tension in the anastomoses.
Patency (primary, primary assisted, secondary, and functional) rates | 6, 12, 18, 24, and 60 months
  Primary patency: defined as the interval between vascular access creation and the first intervention to maintain or restore patency.
  Assisted primary patency: defined as the interval between vascular access creation and the first occlusion (thrombosis), including interventions (operative or endovascular) aimed to maintain the functionality of the vascular access.
  Secondary patency: defined as the interval between vascular access creation and abandonment with or without interventions (operative or endovascular) aimed to maintain or restore the vascular access's functionality Functional patency: defined as an AV access that can be cannulated with two dialysis needles for at least 75% of dialysis sessions within a 4-week period to achieve the prescribed dialysis.
Time to first intervention and to access abandonment | 60 months
Rate of access-related interventions required to achieve/maintain patency | 6, 12, 18, 24, 60 months
Incidence rate of access site infections | 6, 12, 18, 24, and 60 months
  Infections are defined as all device or procedure related infections potentially resulting from surgical manipulations or device cannulation, including both minor and major infections.
Proportion of hemodialysis sessions completed via a central venous catheter (CVC) during the first 12 months of access creation and access cannulation, irrespective of access abandonment | 12 months
Time to the first cannulation | 12 months
  Assessed only in subjects already on dialysis at the time of implant
Following the first cannulation, the number of days with CVC in situ (catheter contact time) during the first 12 months, irrespective of access abandonment | 12 months
Rate of peri-reintervention vascular injuries | 6 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - AKDHC Medical Research Services, LLC, Tuscon, Arizona
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Greenwood Leflore Hospital, Greenwood, Mississippi
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Flow Vascular, Surgery Specialty Hospitals of America, Pasadena, Texas

IPD SHARING:
Plan to Share IPD: No